CLINICAL TRIAL: NCT05897762
Title: The Effects of Telerehabilitation on Upper Extremity Functions and Activities of Daily Living in Chronic Hemiplegic Patients
Brief Title: The Effects of Telerehabilitation in Chronic Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Hacer Karakurt, Student, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HasanKU"
Record Dates: First submitted 2023-02-04; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-03

CONDITIONS: Hemiplegia
Keywords: fuctionallity; chronic hemiplegia; Spastisity; Tele-rehabilitation; upper extremity
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinic Grup (Other): the same exercises were performed in the clinical setting, accompanied by a physiotherapist. The evaluations were made before and after the treatment.
  Interventions: Behavioral: Tele rehabilitation Group

INTERVENTIONS:
Behavioral: Tele rehabilitation Group — It has been determined that the telerehabilitation method applied in chronic hemiplegic patients increases daily living activities, upper extremity functionality, and spasticity levels decrease.

SUMMARY:
The present study was conducted to investigate the effects of telerehabilitation on upper extremity functions and activities of daily living in chronic hemiplegic patients.

DETAILED DESCRIPTION:
A total of 40 chronic hemiplegic subjects were included in the study. The patients were divided into 2 groups by simple randomization method. As the Telerehabilitation Group (TR), Group 1 completed the treatment program, which included upper extremity and lower extremity strengthening exercises, for eight weeks, three days a week for 45-60 minutes, 10 repetitions, with online supervision. Group 2 was planned as a face-to-face training group and the same exercises were performed in the clinical setting, accompanied by a physiotherapist. The evaluations were made before and after the treatment. The Modified Ashworth Scale was used for upper extremity spasticity evaluation. The Wolf Motor Function Test was used to evaluate upper extremity functionality. The Barthel ADL Index was used to evaluate Activities of Daily Living (ADL). The Brunnstrom Staging Survey was used to evaluate the level of motor recovery. The Treatment Satisfaction Inquiry Survey was used to evaluate the satisfaction of the patients with the treatment method. Heart Rate (HR) values and oxygen saturation (SaO2) were measured with Pulse Oximetry to monitor vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with stroke between the ages of 40-70
* It has been 12 months since the stroke
* Individuals with upper extremity spasticity level (Modified Ashworth Scale (MAS) score ≤ 3)
* Hand and upper extremity values above 3 according to Brunnstrom motor staging
* Individuals with ischemic, middle cerebral artery involvement will be taken.

Exclusion Criteria:

* Having advanced apraxia and aphasia
* Patients who do not have the cooperation to perform verbal commands and exercise training
* Patients who have undergone any botulinum toxin application in the last 6 months
* Patients with significant visual and hearing loss
* Individuals who do not have the necessary technological competence to provide remote video communication at home will not be accepted.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
spasticity levels | Pre-Treatment and post treatment evaluations will ve recorded. (8 Weeks periods)
  Spasticty will ve evaluated with Modifiye Ashworth Scale
Upper Extremity functionality | Pre-Treatment and post treatment evaluations will ve recorded. (8 Weeks periods)
  Upper extremity functionality evaluated with DASH

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Kocamaz, Assist Prof, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No